CLINICAL TRIAL: NCT07063758
Title: Biomarker Studies to Predict Treatment Outcomes of Enfortumab Vedotin in Advanced Urothelial Carcinoma
Brief Title: A Biomarker Study to Predict Treatment Outcomes of Enfortumab Vedotin in Advanced Urothelial Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Clinical Trial Center (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital Clinical Trial Center, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Other Study IDs: 202502065RINE
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Advanced Urothelial Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tumor tissue samples and peripheral blood samples (serum) will be retained. Tumor tissues will be used for immunohistochemical analysis of membranous Nectin-4 and ADAM10/17 expression. Serum samples will be collected at predefined time points during treatment to measure soluble Nectin-4 (sNectin-4) levels. Samples may also be used in future biomarker studies, including DNA-based analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EV Therapy Cohort: Patients with advanced urothelial carcinoma who receive enfortumab vedotin-based therapies. Tumor tissue and serum samples will be collected and analyzed for membranous Nectin-4, ADAM10/17, and soluble Nectin-4 (sNectin-4) to assess their association with treatment outcomes.
  Interventions: Other: Biomarker Analysis
- Chemotherapy Cohort: Patients with advanced urothelial carcinoma who receive platinum-based chemotherapy. Tumor tissue and serum samples will be collected and analyzed for membranous Nectin-4, ADAM10/17, and soluble Nectin-4 (sNectin-4) to assess their association with treatment outcomes.
  Interventions: Other: Biomarker Analysis

INTERVENTIONS:
Other: Biomarker Analysis — Tumor tissue and serum samples will be collected and analyzed to evaluate the expression of membranous Nectin-4, ADAM10/17, and levels of soluble Nectin-4 (sNectin-4) as predictive biomarkers in patients with advanced urothelial carcinoma receiving standard therapies.

SUMMARY:
This study aims to find biological markers that help predict how patients with advanced urothelial carcinoma respond to treatment with enfortumab vedotin (EV) or EV-based combination therapies. Since EV can cause significant side effects and is costly, identifying markers such as nectin-4 and related proteins in tumor tissue and blood may help doctors personalize treatment plans. The investigators will enroll about 100 patients receiving EV and compare them to another 100 patients treated with standard chemotherapy. By studying tissue samples and blood at different times, the investigators hope to discover which markers best indicate treatment success or risks. This research could lead to better, safer treatments tailored to each patient's biology.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 y/o
2. Histologically confirmed urothelial carcinoma
3. Radiologically documented locally advanced or metastatic disease
4. Exposure to EV (as monotherapy or in combination with pembrolizumab) or first-line platinum-based chemotherapy
5. Complete and identifiable medical records

Exclusion Criteria:

1. Inadequate or insufficient tumor tissues for analyses
2. Incomplete medical records

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with advanced urothelial carcinoma receiving enfortumab vedotin-based therapies or first-line platinum-based chemotherapy. Participants will be adults aged 20 years or older, of any sex, with available archival tumor tissue and serum samples for biomarker analyses. Patients must have adequate organ function and no prior treatment with enfortumab vedotin.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 months after treatment initiation
  Proportion of patients achieving complete or partial tumor response according to RECIST 1.1 criteria after enfortumab vedotin treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  Time from treatment start to disease progression or death from any cause.
Overall Survival (OS) | Up to 36 months
  Time from treatment initiation to death from any cause.
Treatment-Related Adverse Events | Up to 36 months
  Incidence and severity of adverse events graded by CTCAE v5.0 during treatment.
Association of Nectin-4, ADAM10/17 Expression and Serum Soluble Nectin-4 with Overall Survival, Progression-Free Survival, Objective Response Rate, and Adverse Events | Assessed at baseline and up to 36 months
  To evaluate the correlation between baseline membranous Nectin-4 expression, ADAM10/17 expression (by immunohistochemistry), and serum soluble Nectin-4 levels (by ELISA) with clinical outcomes, including:
  Overall survival (OS)
  Progression-free survival (PFS)
  Objective response rate (ORR) assessed by RECIST v1.1
  Treatment-related adverse events graded by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Jen Hsueh, M.D., Principal Investigator — Department of Medical Oncology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request after publication of the primary results. Data sharing will follow applicable ethical and privacy regulations. Requests can be directed to the Principal Investigator and will require a data use agreement.

REFERENCES:
- [Background] Powles T, Valderrama BP, Gupta S, Bedke J, Kikuchi E, Hoffman-Censits J, Iyer G, Vulsteke C, Park SH, Shin SJ, Castellano D, Fornarini G, Li JR, Gumus M, Mar N, Loriot Y, Flechon A, Duran I, Drakaki A, Narayanan S, Yu X, Gorla S, Homet Moreno B, van der Heijden MS; EV-302 Trial Investigators. Enfortumab Vedotin and Pembrolizumab in Untreated Advanced Urothelial Cancer. N Engl J Med. 2024 Mar 7;390(10):875-888. doi: 10.1056/NEJMoa2312117. PMID 38446675

DOCUMENTS (1):
  • Study Protocol (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT07063758/Prot_000.pdf